CLINICAL TRIAL: NCT03251287
Title: Mechanistic Study of the Effect of Inorganic Sodium Nitrate on Cardiac and Skeletal Muscle Metabolic Efficiency in Patients With Hypertrophic Cardiomyopathy
Brief Title: Nitrite in Hypertrophic Cardiomyopathy (HCM) Study
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of East Anglia (Other)
Collaborators: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other); British Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 201323
Record Dates: First submitted 2017-08-11; First posted 2017-08-16 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-08

CONDITIONS: Cardiomyopathy, Hypertrophic
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — sodium nitrate

STUDY DESIGN:
Intervention Model Description: This is a placebo-controlled, random-order mechanistic study of oral inorganic sodium nitrate versus placebo in cross-over fashion in patients with non obstructive hypertrophic cardiomyopathy and exercise limitation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This will be a double blind study. The placebo and active treatments will appear identical and will be dispensed in identical containers. All trial patients, care providers, outcome assessors and data analysts will remain blind throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium Nitrate (Active Comparator): Following entry into the study, patients will receive a single dose of oral inorganic sodium nitrate (14mmol) on two separate visits, or matching placebo, in random order (i.e. 2x nitrate visits first or 2x placebo visits first) in a cross-over fashion.
  Interventions: Drug: Sodium Nitrate; Diagnostic Test: Phosphorous Magnetic Resonance Spectroscopy; Diagnostic Test: Exercise Stress Transthoracic Echocardiogram
- Placebo (Placebo Comparator): Following entry into the study, patients will receive a single dose of oral inorganic sodium nitrate (14mmol) on two separate visits, or matching placebo, in random order (i.e. 2x nitrate visits first or 2x placebo visits first) in a cross-over fashion.
  Interventions: Drug: Placebo; Diagnostic Test: Phosphorous Magnetic Resonance Spectroscopy; Diagnostic Test: Exercise Stress Transthoracic Echocardiogram

INTERVENTIONS:
Drug: Sodium Nitrate — Single dose of 14mmol oral inorganic sodium nitrate
  Arms: Sodium Nitrate
Drug: Placebo — Single dose of oral matching placebo
  Arms: Placebo
Diagnostic Test: Phosphorous Magnetic Resonance Spectroscopy — On the first visit day of this arm, participants will be lie inside an MRI scanner to take pictures of the heart. The thigh muscle will then be imaged before, during, and after kicking exercises.
Diagnostic Test: Exercise Stress Transthoracic Echocardiogram — On the second visit day of this arm, participants will be asked to lie, semi-erect, on an exercise bed for up to 90 minutes. The echocardiogram will be performed at rest and during peak exercise. The exercise will be in the form of a pedal bike. The exercise levels will be worked out from an upright bicycle exercise test completed by the participants prior to randomization.

SUMMARY:
Inorganic nitrate, which is found at high levels in green leafy vegetables, is reduced to nitrite by bacteria in the mouth, swallowed, and absorbed in the stomach into the blood. Studies have shown that increasing the blood levels of nitrite improves the way that muscles use oxygen and energy during exercise, and potentially blood flow.

Some people (~1 in 500) suffer from a type of genetic heart condition known as hypertrophic cardiomyopathy (HCM). This condition means that the muscle in the heart does not use energy well and becomes larger than average, meaning that they have to tap into the heart's 'energy reserves'. It is not known if nitrite has the same beneficial effects on heart muscle as on other muscles in the body. Our study will explore the mechanism by which nitrite may improve the function and energy status of the heart in HCM.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged between 18 and 80 years.
* Able to provide informed consent.
* Able to understand basic instructions in English.
* A diagnosis of hypertrophic cardiomyopathy based on conventional transthoracic echocardiogram guidelines: left ventricular wall thickness >1.5cm in the absence of sufficient alternative cause.
* Exercise limited by symptoms on exertion (NYHA Class II symptoms or greater).
* PeakVO2 <80% on baseline CPEX.
* The absence of resting LV outflow tract obstruction (peak gradient <30 mm Hg) on TTE.

Exclusion Criteria:

* Significant medical, surgical or psychiatric disease that in the opinion of the patient's attending physician would affect subject safety or influence the study outcome.
* Contraindications for undergoing MRI.
* Hypotension with a systolic blood pressure <90mmHg.
* Severe anaemia with a plasma haemoglobin level <8.0g/dL.
* Known glucose-6-phosphate dehydrogenase (G6PD) deficiency or G6PD deficiency measured at screening in males of African, Asian or Mediterranean decent.
* Female subjects of childbearing potential.
* Haemodynamically significant valve disease.
* Predisposed to acute on chronic limb ischemia evident from a history of claudication or known peripheral arterial disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Cardiac Energetic Status | 3 hours post dose of drug or placebo
  Change in cardiac PCr/ATP ratio on phosphorus MRS between inorganic sodium nitrate and placebo

SECONDARY OUTCOMES:
Skeletal Muscle Mitochondrial Oxidative Capacity/Energetic Status | 3.5 hours post dose of drug or placebo
  Change in PCr recovery half-time on dynamic phosphorus MRS between inorganic sodium nitrate and placebo
Cardiac Diastolic and Systolic Function on exercise | 3 hours post dose of drug or placebo
  Change in measures of diastolic and systolic function on transthoracic echocardiogram at submaximal exercise between inorganic sodium nitrate and placebo
Cardiac Diastolic and Systolic Function at rest | 3 hours post dose of drug or placebo
  Change in measures of diastolic and systolic function on transthoracic echocardiogram at rest between inorganic sodium nitrate and placebo
Plasma levels of Nitrate/Nitrite/NOx | 3 hours post dose of drug or placebo
  Change in blood plasma levels of Nitrate/Nitrite/NOx between inorganic sodium nitrate and placebo

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Frenneaux, MD, Study Chair — University of East Anglia; Sunil V Nair, MD, Principal Investigator — Norfolk and Norwich University Hospitals NHS Foundation Trust
Locations (1):
- Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: No